CLINICAL TRIAL: NCT04351087
Title: Microfragmented Adipose Tissue Versus Platelet-rich Plasma for Knee Osteoarthritis: a Randomized Comparative Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Michael Baria, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019H0448
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Osteoarthritis, Knee; Microfragmented Adipose Tissue; Platelet-Rich Plasma
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Two-treatment parallel-design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Platelet Rich Plasma (Active Comparator): 157cc of whole blood will be harvested via standard venipuncture from the antecubital fossa and mixed with 24cc ACD-A (manufacturer recommends 8cc ACD-A per 52cc of whole blood). 156ml of whole blood will be processed in the FDA Cleared Angel cPRP system at 2% hematocrit. 1ml of whole blood and the resultant PRP will be analyzed in the Sysmex XN-350 for complete analysis (platelet, leukocyte, red blood cell counts). The remaining PRP will be injected under sterile technique using ultrasound-guidance through a superolateral approach. For patient comfort, 2cc of 1% lidocaine can be administered using a 26-gauge needle (into soft tissues only). PRP will then be injected using a 25-guage needle. A maximum of 6ml of PRP will be injected. Injection site will be cleaned and bandaged and patient will be dismissed with post-injection precautions and 1 month follow-up scheduled.
  Interventions: Device: Platelet Rich Plasma
- Microfragmented adipose tissue (Active Comparator): Adipose is aspirated from the subcutaneous tissue of the buttock or abdomen. Aspiration site is injected with 10ml 1% lidocaine with epinephrine. A small poke incision is made with an 11-blade scalpel. Then 120ml of Klein solution is injected into the adipose tissue. Solution sits for 15 minutes to allow for adequate anesthesia. Aspiration cannula is inserted and moved in a back and forth motion for 2 minutes to allow for adipose aspiration. 30ml fat will be aspirated. Aspiration site is cleaned and bandaged. The aspirated fat is processed using the Lipogems system. 30ml of adipose is transferred to the device, saline is run through the device to remove oils and then approximately 5-7ml of adipose tissue is removed and ready for injection. The Microfragmented adipose tissue are then injected in identical fashion to the PRP above.
  Interventions: Device: Platelet Rich Plasma

INTERVENTIONS:
Device: Platelet Rich Plasma — Platelet rich plasma: 157cc of whole blood will be collected, processed, and injected into the knee joint under sterile technique using ultrasound-guidance.
  Microfragmented adipose tissue: Adipose will be aspirated from the subcutaneous tissue of the buttock or abdomen, processed, and injected into the knee joint under sterile technique using ultrasound-guidance.
  Other Names: Microfragmented adipose tissue

SUMMARY:
The study aims to conduct a randomized trial comparing the clinical outcomes of PRP (standard intervention) versus Microfragmented adipose tissue (investigational) for the treatment of knee osteoarthritis.

Hypothesis: Both interventions will result in significant improvement in patient-reported outcomes. We hypothesize that Microfragmented adipose tissue will provide superior outcomes.

DETAILED DESCRIPTION:
Background

Knee osteoarthritis is a leading cause of disability worldwide. Standard of care treatments for knee OA include activity modification, weight loss, therapeutic exercise and injections like corticosteroids and viscosupplement. These commonly used non-operative treatments focus on symptom palliation, but are not disease modifying.

Orthobiologics have emerged as a promising treatment for knee OA. The most widely studied orthobiologic is platelet-rich plasma (PRP). PRP is a dense concentration of platelets derived from autologous whole blood and platelets are concentrated 2-5x compared to baseline. The platelets have demonstrated anti-inflammatory and chondroprotective properties.6 PRP has been shown superior to placebo and viscosupplement for knee OA in several clinical trials.

While PRP is the most widely studied and used orthobiologic, it contains only platelets. Therefore, a simple, office-based intervention able to collect additional reparative cells to treat knee OA would be ideal. Adipose (fat) is a known source of reparative cells like pericytes and it can be easily and safely aspirated in the clinic. The adipose tissue aspiration and processing is accomplished through a simple process. After local anesthesia to the site of adipose aspiration (lower abdomen or buttock), 30ml of adipose is aspirated through a cannula. That adipose is then processed in accordance with FDA guidelines including minimal manipulation to remove oils.. Using minimally manipulated Microfragmented adipose tissue has been shown safe for use as injection therapy for knee OA for 3 years.

Methods:

Patients / Outcome Measures / Sample size: Patients with unilateral symptomatic knee OA will be recruited from the sports medicine and orthopedics clinics, as well as advertising flyers within the clinic. All patients' first visit will include a medical evaluation and assess best treatment plan for that patient, regardless of candidacy for this study. This evaluation includes x-rays of their knees as a standard part of the evaluation. If they meet criteria and choose to enroll, they will be randomly assigned to either the PRP or Microfragmented adipose tissuetreatment group. Patients will complete follow up visits and surveys at defined time points through 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-75 years
* BMI < 40
* Diagnosis of knee OA (primary and post-traumatic)
* Radiographic evidence of OA of the target knee (Kellgren-Lawrence grades 1-4)
* Continued OA pain in the target knee despite at least 6 weeks of 1 of the following nonoperative treatments: activity modification, weight loss attempt, physical therapy, or NSAID / acetaminophen.
* Knee Osteoarthritis Outcomes Score (KOOS)-Pain subscale 20-65
* Working knowledge of English language (to be able to complete all outcome scores)
* Ability to attend all follow-up appointments

Exclusion Criteria:

* Isolated patellofemoral OA
* 3+ effusion of the target knee (stroke test grading system)
* Significant (10 degree) valgus or varus deformities
* Prior injection therapy:
* Steroid injection in target knee in the last 3 months
* Viscosupplementation in target knee in the last 6 months
* PRP in the target knee in the last 1 year
* No other cellular treatments in index knee (bone marrow, amniotic suspensions etc) all time
* Participation in any experimental device or drug study within 1 year before screening visit
* Oral or IM steroids for last 3 months
* Medical condition that may impact outcomes of procedure including:
* anemia
* thrombocytopenia
* bleeding disorders
* inflammatory disorders like rheumatoid arthritis, lupus
* diabetes
* any history of cancer (other than non-melanoma skin malignancies)
* taking anticoagulants (aspirin, Plavix, eliquis, Xarelto, warfarin, lovenox)
* Taking immunosuppressants, having a severe systemic infection
* Previous cartilage repair procedure on the injured cartilage surface (ie, OATS, ACI, MFX)
* Previous surgery at the target knee within the past 1 year
* Any degree of cognitive impairment.
* OA of either hip
* Pregnancy, lactating, or intent to become pregnant during treatment period
* Gout
* History of infection or current infection at the affected joint
* Smoking

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Baria, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Sports Medicine Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1323-30. doi: 10.1136/annrheumdis-2013-204763. Epub 2014 Feb 19. PMID 24553908
- [Background] Hermann W, Lambova S, Muller-Ladner U. Current Treatment Options for Osteoarthritis. Curr Rheumatol Rev. 2018;14(2):108-116. doi: 10.2174/1573397113666170829155149. PMID 28875826
- [Background] Liu Q, Niu J, Huang J, Ke Y, Tang X, Wu X, Li R, Li H, Zhi X, Wang K, Zhang Y, Lin J. Knee osteoarthritis and all-cause mortality: the Wuchuan Osteoarthritis Study. Osteoarthritis Cartilage. 2015 Jul;23(7):1154-7. doi: 10.1016/j.joca.2015.03.021. Epub 2015 Mar 25. PMID 25819581
- [Background] Dai WL, Zhou AG, Zhang H, Zhang J. Efficacy of Platelet-Rich Plasma in the Treatment of Knee Osteoarthritis: A Meta-analysis of Randomized Controlled Trials. Arthroscopy. 2017 Mar;33(3):659-670.e1. doi: 10.1016/j.arthro.2016.09.024. Epub 2016 Dec 22. PMID 28012636
- [Background] Marx RE. Platelet-rich plasma (PRP): what is PRP and what is not PRP? Implant Dent. 2001;10(4):225-8. doi: 10.1097/00008505-200110000-00002. No abstract available. PMID 11813662
- [Background] Moussa M, Lajeunesse D, Hilal G, El Atat O, Haykal G, Serhal R, Chalhoub A, Khalil C, Alaaeddine N. Platelet rich plasma (PRP) induces chondroprotection via increasing autophagy, anti-inflammatory markers, and decreasing apoptosis in human osteoarthritic cartilage. Exp Cell Res. 2017 Mar 1;352(1):146-156. doi: 10.1016/j.yexcr.2017.02.012. Epub 2017 Feb 13. PMID 28202394
- [Background] Cole BJ, Karas V, Hussey K, Pilz K, Fortier LA. Hyaluronic Acid Versus Platelet-Rich Plasma: A Prospective, Double-Blind Randomized Controlled Trial Comparing Clinical Outcomes and Effects on Intra-articular Biology for the Treatment of Knee Osteoarthritis. Am J Sports Med. 2017 Feb;45(2):339-346. doi: 10.1177/0363546516665809. Epub 2016 Oct 21. PMID 28146403
- [Background] Gormeli G, Gormeli CA, Ataoglu B, Colak C, Aslanturk O, Ertem K. Multiple PRP injections are more effective than single injections and hyaluronic acid in knees with early osteoarthritis: a randomized, double-blind, placebo-controlled trial. Knee Surg Sports Traumatol Arthrosc. 2017 Mar;25(3):958-965. doi: 10.1007/s00167-015-3705-6. Epub 2015 Aug 2. PMID 26233594
- [Background] Sanchez M, Fiz N, Azofra J, Usabiaga J, Aduriz Recalde E, Garcia Gutierrez A, Albillos J, Garate R, Aguirre JJ, Padilla S, Orive G, Anitua E. A randomized clinical trial evaluating plasma rich in growth factors (PRGF-Endoret) versus hyaluronic acid in the short-term treatment of symptomatic knee osteoarthritis. Arthroscopy. 2012 Aug;28(8):1070-8. doi: 10.1016/j.arthro.2012.05.011. PMID 22840987
- [Background] Smith PA. Intra-articular Autologous Conditioned Plasma Injections Provide Safe and Efficacious Treatment for Knee Osteoarthritis: An FDA-Sanctioned, Randomized, Double-blind, Placebo-controlled Clinical Trial. Am J Sports Med. 2016 Apr;44(4):884-91. doi: 10.1177/0363546515624678. Epub 2016 Feb 1. PMID 26831629
- [Background] De Francesco F, Ricci G, D'Andrea F, Nicoletti GF, Ferraro GA. Human Adipose Stem Cells: From Bench to Bedside. Tissue Eng Part B Rev. 2015 Dec;21(6):572-84. doi: 10.1089/ten.TEB.2014.0608. Epub 2015 Jun 17. PMID 25953464
- [Background] Dragoo JL, Chang W. Arthroscopic Harvest of Adipose-Derived Mesenchymal Stem Cells From the Infrapatellar Fat Pad. Am J Sports Med. 2017 Nov;45(13):3119-3127. doi: 10.1177/0363546517719454. Epub 2017 Aug 17. PMID 28816507
- [Background] Russo A, Condello V, Madonna V, Guerriero M, Zorzi C. Autologous and micro-fragmented adipose tissue for the treatment of diffuse degenerative knee osteoarthritis. J Exp Orthop. 2017 Oct 3;4(1):33. doi: 10.1186/s40634-017-0108-2. PMID 28975547
- [Background] Russo A, Screpis D, Di Donato SL, Bonetti S, Piovan G, Zorzi C. Autologous micro-fragmented adipose tissue for the treatment of diffuse degenerative knee osteoarthritis: an update at 3 year follow-up. J Exp Orthop. 2018 Dec 19;5(1):52. doi: 10.1186/s40634-018-0169-x. PMID 30569417
- [Derived] Baria M, Barker T, Durgam S, Pedroza A, Flanigan D, Jia L, Kaeding C, Magnussen R. Microfragmented Adipose Tissue Is Equivalent to Platelet-Rich Plasma for Knee Osteoarthritis at 12 Months Posttreatment: A Randomized Controlled Trial. Orthop J Sports Med. 2024 Mar 18;12(3):23259671241233916. doi: 10.1177/23259671241233916. eCollection 2024 Mar. PMID 38510323
- [Derived] Baria M, Pedroza A, Kaeding C, Durgam S, Duerr R, Flanigan D, Borchers J, Magnussen R. Platelet-Rich Plasma Versus Microfragmented Adipose Tissue for Knee Osteoarthritis: A Randomized Controlled Trial. Orthop J Sports Med. 2022 Sep 16;10(9):23259671221120678. doi: 10.1177/23259671221120678. eCollection 2022 Sep. PMID 36147791

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 8 participants were excluded prior to intervention due to not meeting inclusion criteria.
Groups:
- Platelet Rich Plasma: 157cc of whole blood will be harvested via standard venipuncture from the antecubital fossa and mixed with 24cc ACD-A (manufacturer recommends 8cc ACD-A per 52cc of whole blood). 156ml of whole blood will be processed in the FDA Cleared Angel cPRP system at 2% hematocrit. 1ml of whole blood and the resultant PRP will be analyzed in the Sysmex XN-350 for complete analysis (platelet, leukocyte, red blood cell counts). The remaining PRP will be injected under sterile technique using ultrasound-guidance through a superolateral approach. For patient comfort, 2cc of 1% lidocaine can be administered using a 26-gauge needle (into soft tissues only). PRP will then be injected using a 25-guage needle. A maximum of 6ml of PRP will be injected. Injection site will be cleaned and bandaged and patient will be dismissed with post-injection precautions and 1 month follow-up scheduled.
  Platelet Rich Plasma: Platelet rich plasma: 157cc of whole blood will be collected, processed, and injected into the knee joint under sterile technique using ultrasound-guidance.
  Microfragmented adipose tissue: Adipose will be aspirated from the subcutaneous tissue of the buttock or abdomen, processed, and injected into the knee joint under sterile technique using ultrasound-guidance.
- Microfragmented Adipose Tissue: Adipose is aspirated from the subcutaneous tissue of the buttock or abdomen. Aspiration site is injected with 10ml 1% lidocaine with epinephrine. A small poke incision is made with an 11-blade scalpel. Then 120ml of Klein solution is injected into the adipose tissue. Solution sits for 15 minutes to allow for adequate anesthesia. Aspiration cannula is inserted and moved in a back and forth motion for 2 minutes to allow for adipose aspiration. 30ml fat will be aspirated. Aspiration site is cleaned and bandaged. The aspirated fat is processed using the Lipogems system. 30ml of adipose is transferred to the device, saline is run through the device to remove oils and then approximately 5-7ml of adipose tissue is removed and ready for injection. The Microfragmented adipose tissue are then injected in identical fashion to the PRP above.
  Platelet Rich Plasma: Platelet rich plasma: 157cc of whole blood will be collected, processed, and injected into the knee joint under sterile technique using ultrasound-guidance.
  Microfragmented adipose tissue: Adipose will be aspirated from the subcutaneous tissue of the buttock or abdomen, processed, and injected into the knee joint under sterile technique using ultrasound-guidance.
Period: Overall Study
Arm/Group | Platelet Rich Plasma | Microfragmented Adipose Tissue
Started | 36 | 35
Completed | 23 | 26
Not Completed | 13 | 9
Not completed — Lost to Follow-up | 7 | 3
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lack of Efficacy | 3 | 2

BASELINE CHARACTERISTICS:
Population: 8 were excluded prior to randomization due to not meeting inclusion criteria. 36 prp and 35 microfragmented adipose tissue (MFAT) were randomized. 3 prp and 4 MFAT participants withdrew before intervention 7 prp and 3 MFAT were lost to follow up, and 3 PRP and 2 MFAT discontinued follow up after receiving intervention. That left 23 PRP and 26 MFAT for statistical analysis on baseline and 1 year outcomes.
Groups:
- Total: Total of all reporting groups
Arm/Group | Platelet Rich Plasma | Microfragmented Adipose Tissue | Total
Number analyzed (Participants) | 23 | 26 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Demographics were analyzed on the cohort that completed enrollment.
  years | 52.8 (14.0) | 56.7 (7.8) | 56.3 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Demographics were analyzed on the cohort that completed enrollment.
  Participants
    Female | 7 | 18 | 25
    Male | 16 | 8 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Demographics were analyzed on the cohort that completed enrollment.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 2 | 1 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 4 | 3 | 7
    White | 17 | 22 | 39
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Knee Injury and Osteoarthritis Outcome Pain Score [KOOS Pain] [Mean (Standard Deviation); unit: units on a scale] — The Knee injury and Osteoarthritis Outcome Pain Score [KOOS questionnaire] is a self-reported outcome measure assessing the patient's opinion about the pain in their knee. Standardized answer options are given [5 Likert boxes] and each question is assigned a score from 0 to 4. A normalized score [100 indicating no pain and 0 indicating extreme pain] is calculated. Population: Measure Analysis Population Description: Demographics were analyzed on the cohort that completed enrollment.
  units on a scale | 51.7 (10.8) | 51.1 (10.2) | 51.4 (10.3)

OUTCOME MEASURES:

1. Primary Outcome: KOOS Pain [Knee Injury and Osteoarthritis Outcome Score]
Description: The Knee injury and Osteoarthritis Outcome Pain Score [KOOS questionnaire] is a self-reported outcome measure assessing the patient's opinion about the pain in their knee. Standardized answer options are given [5 Likert boxes] and each question is assigned a score from 0 to 4. A normalized score [100 indicating no pain and 0 indicating extreme pain] is calculated.
Time Frame: 6 months
Population: Out of 36 subjects randomized to receive platelet rich plasma, 33 received allocated intervention and 3 voluntarily withdrew prior to intervention. Out of the 33, 7 were lost to follow up and 3 discontinued intervention. Out of 35 subjects randomized to receive microfragmented adipose tissue, 31 received allocated intervention and 4 voluntarily withdrew prior to intervention. Out of the 31, 3 were lost to follow up and 2 discontinued intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Platelet Rich Plasma | Microfragmented Adipose Tissue
Number analyzed (Participants) | 23 | 26
units on a scale | 79.95 (17.86) | 77.78 (19.33)
Statistical Analysis 1: Comparison: Platelet Rich Plasma vs Microfragmented Adipose Tissue; Test type: Equivalence — Power analysis based on (MCID) for the KOOS-Pain, alpha 0.05 & SD 15 points, 88 patients (44/group) would be required to detect a 9-point difference between treatment groups with 80% power. Due to change in regulatory requirements during accrual, enrollment was halted at 79 patients with 71 meeting inclusion criteria. A repeated power calculation demonstrated that the study achieved 56% power to detect a between-group difference in excess of the 9-point MCID for the KOOS-Pain; p = 0.69, t-test, 2 sided; Mean Difference (Final Values) = 2.17, 95% CI 2-sided [-8.57 to 12.92]

2. Secondary Outcome: VAS [Visual Analog Pain Scale] Pain Score
Description: The visual analog pain scale [VAS] is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between 0 [no pain] and 10 [worst pain].
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Platelet Rich Plasma | Microfragmented Adipose Tissue
Number analyzed (Participants) | 23 | 26
units on a scale | 1.6 (0.4) | 1.4 (0.4)

3. Secondary Outcome: Tegner Activity Scale
Description: The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Platelet Rich Plasma | Microfragmented Adipose Tissue
Number analyzed (Participants) | 23 | 26
score on a scale | 3.9 (0.3) | 4.3 (0.3)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from baseline through 1 year post injection.
Arm/Group | Platelet Rich Plasma | Microfragmented Adipose Tissue
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/35
Other Adverse Events (participants affected / at risk) | 11/36 | 8/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Platelet Rich Plasma (N=36) | Microfragmented Adipose Tissue (N=35)
Swelling (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT04351087/Prot_SAP_002.pdf
  • Informed Consent Form (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT04351087/ICF_003.pdf